CLINICAL TRIAL: NCT00117026
Title: Can Oral Benfotiamine Supplementation Influence Progression of Microvascular Complications in Patients With Type 1 Diabetes?
Brief Title: Effects of Vitamin B1 in Type 1 Diabetic Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital, Aker (Other)
Collaborators: The Research Council of Norway (Other)
Responsible Party: Principal Investigator, Kristian F. Hanssen, Professor, Oslo University Hospital
Organization: Oslo University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AkerU
Record Dates: First submitted 2005-06-30; First posted 2005-07-04 (Estimated); Last update posted 2013-05-10 (Estimated); Status verified 2013-05

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Diabetes Complications; benfotiamine; type 1 diabetes; elevated urinary albumin excretion; nerve function; advanced glycation end products
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Complications | interventions — benphothiamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Benfotiamine (Experimental): Benfotiamine 300mg/day
  Interventions: Drug: Benfotiamine
- Placebo (Placebo Comparator): Placebo for benfotiamine
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Placebo for benfotiamine
  Arms: Placebo
Drug: Benfotiamine — 300mg/day
  Other Names: S-benzoylthiamine O-monophoshate
  Arms: Benfotiamine

SUMMARY:
The purpose of this study is to determine whether benfotiamine supplementation can reduce markers of microvascular complications in type 1 diabetic patients.

DETAILED DESCRIPTION:
Despite intensive strategies designed to achieve good metabolic control, diabetic patients are still at a markedly increased risk of eye and kidney disease, nerve damage, limb amputation, stroke and myocardial infarction as a result of long-term hyperglycemia. It has recently been shown that supplementation with lipid soluble vitamin B1 (benfotiamine) in diabetic rats could effectively block three major biochemical pathways of hyperglycemic damage. It has also been shown that supplementation prevented the development of experimental diabetic retinopathy and nephropathy, without changes in glycemic control. However, the applicability of the above findings to humans is unknown, and the diabetic late complications in experimental animals do not in every aspect mirror the human diabetic complications.

This project will allow us to evaluate the potential of benfotiamine to reduce or prevent the further development of microvascular disease in type 1 diabetics.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes (of at least 15 years duration) as assessed by medical history.

Exclusion Criteria:

* Macroalbuminuria
* Symptomatic gastroparesis. Diabetic nephropathy with a creatinine clearance less than 60 cc/min.
* Evidence of chronic infection.
* History of any malignancy.
* Any chronic medical condition that unduly increases the risk for the potential enrollee as judged by study investigators.
* Pregnancy, breastfeeding or planned pregnancy within two years.
* Supplementation with thiamine > 2mg per day and/or alpha-lipoic acid
* Chronic alcoholism/alcohol abuse.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2005-08; Primary Completion 2010-06 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Lower-limb nerve conduction velocity | 24 months

SECONDARY OUTCOMES:
Serum advanced glycation end products (AGEs) and markers of inflammation (CRP, IL-6, VCAM-1) | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Kristian F Hanssen, MD, PhD, Principal Investigator — University Hospital, Aker
Locations (1):
- Aker University Hospital, Oslo, Norway

REFERENCES:
- [Derived] Fraser DA, Diep LM, Hovden IA, Nilsen KB, Sveen KA, Seljeflot I, Hanssen KF. The effects of long-term oral benfotiamine supplementation on peripheral nerve function and inflammatory markers in patients with type 1 diabetes: a 24-month, double-blind, randomized, placebo-controlled trial. Diabetes Care. 2012 May;35(5):1095-7. doi: 10.2337/dc11-1895. Epub 2012 Mar 23. PMID 22446172